CLINICAL TRIAL: NCT04942808
Title: A Comparative Observational Study of the Crestal Bone Loss Around Bone Level Versus Tissue Level Implants in Non-compliant Patients With Healthy or Reduced Periodontium After 5-8 Years in Function"
Brief Title: A Study of the Crestal Bone Loss Around Bone Level Versus Tissue Level Implants in Non-compliant Patients With Healthy or Reduced Periodontium After 5-8 Years in Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Layal Bou Semaan, Resident, Saint-Joseph University
Other Study IDs: FMDA9/21
Record Dates: First submitted 2021-06-16; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Periimplantitis; Marginal Bone Loss
Keywords: Oral hygiene; Dental implant; Periodontal maintenance; Marginal bone loss; Tissue level implant; Bone level implant; Internal connection; External connection
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Periapical radiographs — Periapical radiographs on reevaluation

SUMMARY:
The goal is to evaluate, after 5 to 8 years, the marginal bone loss around tissue-level implants and bone-level implants in patients who have not followed the maintenance program.

Medical records of patients who have been implanted for at least 5 to 8 years and who have been lost during this period are collected from three private clinics in Beirut,Lebanon and the Saint Joseph University Health Center in Beirut,Lebanon.

On an individual sheet, the patient as well as the implants data will be noted. Patients will be called for reevaluation after 5-8 years. After signing the informed consent, the measurements by a PCP-15 probe of the plaque index (FMPS) and the bleeding index (FMBS) as well as the height of the keratinized tissue are indicated on the sheet. If the smoking status has changed, this will be mentioned too.

The marginal bone loss will be measured on the X-rays taken immediately after the implant placement, after 1 year of loading and then at the reevaluation session.

DETAILED DESCRIPTION:
On the individual sheet for each patient, the data concerning the name, age, sex, general condition, smoking status, periodontal status , the number of follow-up sessions and the plaque index as well as bleeding on probing (if noted in the file before placing the implants) will be recorded.

Then, the data concerning the implant such as the site (maxilla or mandibular), the type of implant, the length, the diameter, the surface, sealed or screwed, presence of a cantilever, hiatus or over-contour, a one or two surgical time, the date of placement and the number of years of operation will also be noted on the form.

Patients will be called for reassessment appointments after 5-8 years. After signing the informed consent, the measurements by a PCP-15 periodontal probe of the plaque index (FMPS), bleeding on probing (FMBS) as well as the height and thickness of the keratinized mucosa are indicated on the sheet. The smoking status will also be updated and indicated.

Implants will be classified into one of these groups:

1. Patients with tissue implants (TL).
2. Patients with bone level implants with internal connection (BL, Internal hex).
3. Patients with bone level implants with external connection (BL, External hex).

X-rays taken after insertion, after 1 year of loading and after 5-8 years will be collected and analyzed on the DBSWIN software. Mesial and distal bone loss after implant placement and after 5 to 8 years will be measured on retro-alveolar radiographs with calibration and recorded on the patient file. The total bone loss will then be calculated.

The radiographic measurement technique is as follows. The platform of the mesial and distal implant (MIS: Mesial Implant Shoulder and DIS: Distal Implant Shoulder) will be defined and a line (A) connecting the two is drawn. Another line (B) tangential to the apex of the implant and parallel to A is also drawn. The bisecting line at A and B is therefore produced and measured to assess the distorted implant length (DIL: Distorted Implant Length). Bone level (BL) measurements will be recorded from the implant platform (MIS-DIS) to the most coronary bone-to-implant contact (BIC) on the mesial and distal sides of each implant. The length of the implant will be used as an actual measurement to calibrate the other measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone the initial phase followed by implant placement in the posterior region.
* Implants placed for more than 5 years.
* The implant systems selected are:

  * Tissue Level Implants: Straumann (Straumann Dental Implants System, Switzerland),
  * Bone Level implants: Branemark, 3i Biomet (external and internal connection), Nobel replace and Astra.
* Patients who did not comply with the maintenance program and who missed more than 30% of appointments.

Exclusion Criteria:

* Systemic diseases (uncontrolled diabetes, drugs which may affect bone metabolism).
* Totally edentulous.
* Severe periodontitis not stabilized
* Inappropriate, unavailable or distorted x-rays.
* Augmented sites.
* Implants placed at a supra or infraosseous level.
* Implants placed immediately after extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who had implants between 2012 and 2015 and who did not follow a maintenance program and whose inclusion criteria are present will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-29 (Estimated); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | 5 to 8 years
  It will be measured mesially and distally on each implant platform until the bone's first coronal contact with the implant. Then, the total bone loss on each implant will be calculated. This is done on the software in millimeters.
Level of oral hygiene | 5 to 8 years
  The second factor studied is the level of hygiene which will be calculated by measuring the plaque index and bleeding on probing. This is done with a PCP-15 periodontal probe by a light sweeping movement at the level of the 4 sites of each tooth and implant and then written on the personalized card for each patient.

SECONDARY OUTCOMES:
Smoking status | 5 to 8 years
  Non-smoker, smoker <10 cig/d, smoker equal or > to 10 cig/d, Former smoker
Periodontal status | 5 to 8 years
  Gingivitis or periodontitis with stage and grade
success and survival of the implant | 5 to 8 years
  1) absence of persistent pain, dysesthesia or paresthesia 2) absence of peri-implant infection with or without suppuration 3) absence of noticeable mobility of the implant and 4) absence of persistent peri-implant bone resorption> 1.5 mm during the first year of loading and 0.2 mm per year for the following years.
Years in function | 5 to 8 years
  Years in function
Height and thickness of the peri-implant keratinized mucosa | 5 to 8 years
  Height and thickness of the peri-implant keratinized mucosa
Overhang or hiatus or cantilever | 5 to 8 years
  Overhang or hiatus or cantilever
Full mouth plaque score | 1 year
  With a periodontal probe, we measure at 4 sites (vestibular, mesial, distal, palatine / lingual) of each implant and tooth, we note 0 / - in the absence of plaque and 1 / + in the presence of plaque.
Full mouth bleeding score | 1 year
  With a periodontal probe and after a gentle sweeping motion over the marginal surface of the implant, detect the presence or absence of bleeding at the 4 sites of each implant and tooth denoted by 1 / + and 0 / - respectively.

OTHER OUTCOMES:
Implant position | 5 to 8 years
  Maxilla or Mandible
Type of prosthesis | 5 to 8 years
  screwed or sealed
Surgical times | 5 to 8 years
  One or two
Number of implants | 5 to 8 years
  Multiple or unitary
Implant surface | 5 to 8 years
  The implant surface is usually related to the implant type indicated in the patient file

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University of Beirut, Beirut, Mount Lebanon, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF